CLINICAL TRIAL: NCT06111703
Title: Knowledge, Attitude and Practice in Utilization of Vital Pulp Therapy in Permanent Teeth by Pediatric Dentists in Egypt: A Cross-sectional Study
Brief Title: Knowledge, Attitude and Practice in Utilization of Vital Pulp Therapy in Permanent Teeth by Pediatric Dentists in Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Maher Gindy, Resident in pediatric dentistry department at Misr International University, Cairo University
Other Study IDs: 1996
Record Dates: First submitted 2023-10-21; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Vital Pulp Therapy
Keywords: Vital Pulp Therapy; Permanent Teeth; Pediatric Dentists

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Knowledge assessment — Knowledge, Attitude and Practice Survey

SUMMARY:
Conducting this questionnaire will help in collecting information about the extent of knowledge, attitude, and practice of utilization of vital pulp therapy in permanent teeth among pediatric dentists in Egypt. This will aid in identifying the knowledge gap, interest, attitude, and practice challenges regarding vital pulp therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric dentists who work in Egypt.
* Dentists who finished any postgraduate study in pediatric dentistry.
* The workplace should be anywhere in Egypt

Exclusion Criteria:

* Dentists who did not practice for the last 5 years.
* Responses with incomplete information

Ages: 24 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pediatric Dentists in Egypt
Sampling Method: Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Vital Pulp Therapy in Permanent Teeth | From the 1st of December- 2023, to the 29th of February- 2024.
  Measured by a KAP questionnaire, and the measuring unit is multiple choice questions.

SECONDARY OUTCOMES:
Attitude and Practice towards Vital Pulp Therapy in Permanent Teeth | From the 1st of December- 2023, to the 29th of February- 2024.
  Measured by a KAP questionnaire, and the measuring unit is multiple choice questions.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bogen G, Dammaschke T, Chandler N. Vital pulp therapy. In: Berman L, Hargreaves KM, editors. Pathways of the Pulp. 12th ed. St. Louis, MO: Elsevier; 2021.
- [Background] Guan X, Zhou Y, Yang Q, Zhu T, Chen X, Deng S, Zhang D. Vital Pulp Therapy in Permanent Teeth with Irreversible Pulpitis Caused by Caries: A Prospective Cohort Study. J Pers Med. 2021 Nov 1;11(11):1125. doi: 10.3390/jpm11111125. PMID 34834477
- [Background] Parmar G, Singh S, Hegde JA, Kumar M, Kalyan S. Launching a new fellowship in microrestorative and endodontics for postgraduates in conservative dentistry and endodontics. J Conserv Dent. 2020 Jul-Aug;23(4):370-373. doi: 10.4103/JCD.JCD_328_20. Epub 2021 Jan 16. PMID 33623238
- [Background] Wisniewski JF, Norooz S, Callahan D, Mohajeri A. Survey of Vital Pulp Therapy Treatment in Permanent Dentition Being Taught at U.S. Dental Schools. J Endod. 2022 Sep;48(9):1107-1112. doi: 10.1016/j.joen.2022.06.009. Epub 2022 Jul 5. PMID 35798124
- [Background] Kakudate N, Yokoyama Y, Sumida F, Matsumoto Y, Gordan VV, Gilbert GH. Dentists' practice patterns of treatment for deep occlusal caries: Findings from a dental practice-based research network. J Dent. 2019 May;84:76-80. doi: 10.1016/j.jdent.2019.03.009. Epub 2019 Mar 29. PMID 30935965
- [Background] Doumani MD, Arnous WA, Alsafadi MF, Alnazer HA, Alanazi SM, Alotaibi KS, Al-Ammari AI. The Vital Pulp Therapy of Permanent Teeth: A Dental Practitioner's Perspective from Saudi Arabia. J Int Soc Prev Community Dent. 2020 Jun 15;10(3):300-308. doi: 10.4103/jispcd.JISPCD_69_19. eCollection 2020 May-Jun. PMID 32802776
- [Result] AAE Position Statement on Vital Pulp Therapy. J Endod. 2021 Sep;47(9):1340-1344. doi: 10.1016/j.joen.2021.07.015. Epub 2021 Aug 3. No abstract available. PMID 34352305
- [Result] American Academy of Pediatric Dentistry. Pulp therapy for primary and immature permanent teeth. The Reference Manual of Pediatric Dentistry. Chicago, Ill.: American Academy of Pediatric Dentistry; 2022:415-23.